CLINICAL TRIAL: NCT00686894
Title: Study of Peripheral Enthesitis With Ultra Sonography Doppler in Spondyloarthropathies Treated With Infliximab
Brief Title: Enthesitis With Ultra Sonography Doppler in Spondyloarthropathies Treated With Infliximab (Study P04440)
Acronym: EUSpA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor Enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P04440; 2006-001579-40
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2010-03-05 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Spondylitis, Ankylosing; SpA
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infliximab 5 mg/kg (Experimental): Infliximab infusions: 5 mg/kg at weeks 0, 2, and 6.
  Interventions: Procedure: PDUS; Drug: Infliximab

INTERVENTIONS:
Procedure: PDUS — PDUS scored for each enthesitis every 2 weeks for 24 weeks.
Drug: Infliximab — * 5 mg/kg
  * IV
  * Frequency : weeks 0,2,6
  Other Names: SCH 215596; REMICADE

SUMMARY:
Subjects will be given 3 infusions of infliximab according to the label at week 0, 2, and 6. Subjects will be followed for a maximum of 18 weeks or until relapse. This study will assess the ability of the Power Doppler Ultrasonography (PDUS) to be a reliable marker of enthesitis response and relapse in subjects treated with infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate willingness to participate in study, adhere to dose and visit schedules, and comply with procedures by signing a written informed consent.
* Negative serum pregnancy test at Week 0.
* Men and women over 18 years of either sex and any race.
* Free of any clinically relevant disease other than SpA that would in the principal investigator's and/or sponsor's opinion, interfere with the conduct of study or its evaluations.
* Eligible for anti-tumor necrosis factor (TNF) treatment according to applicable local guidelines.
* Fulfill the following criteria: European Spondyloarthropathy Study group (ESSG) Classification Criteria, and/or Amor Criteria, and/or New York modified criteria.
* Disease duration of SpA >6 months.
* Incomplete response to non-steriodal anti-inflammatory drug (NSAID).
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) >4 including item 2 (axial pain) >=3 on a scale from 0 to 10.
* At least 1 enthesitis assessed by PDUS.
* C-reactive protein (CRP) twice upper normal laboratory value or inflammatory signal on magnetic resonance imaging (MRI) of spine or sacroiliac joint within the last 3 months.
* Practicing adequate contraception during the study and for 6 months after last infusion.
* Week 0 laboratory tests must meet protocol criteria.

Exclusion Criteria:

* Is a female who is pregnant, or intends to become pregnant during the study (or within 6 months after receiving the last infusion);
* Is a female who is nursing, or intends to be nursing during the study or within 6 month after having received the last infusion;
* Has childbearing potential without contraception throughout the study and for 6 months after receiving the last infusion.
* Has not observed the designated washout periods for any of the prohibited medications outlined in the protocol;
* Has any clinically significant deviation from the appropriate reference range in the physical examination, Chest X-ray, that, in the investigator's judgment, may interfere with the study evaluation or affect subject safety;
* Is in a situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Is on the staff, affiliated with, or a family member of the staff personnel directly involved with this study;
* Is allergic to or has sensitivity to the study drug or its excipients;
* Has intolerance to or contraindication for infliximab.
* Has an history of allergy to murine products.
* Is uncooperative or has not signed the consent form.
* Cannot understand the protocol.
* Has participated in a study within 3 months prior to inclusion.
* Had treatment with unstable doses of analgesic drugs (paracetamol, phenylbutazone, morphine) steroid, NSAID, or immunosuppressive agent, including methotrexate, within 4 weeks prior to inclusion.
* Had Intra articular steroid within 4 weeks prior to inclusion.
* Had Previous treatment with infliximab
* Had previous treatment with etanercept, adalimumab or any other TNF agent within 2 last months.
* Had an history of, ongoing or recurrent medical condition as follows :

  * Infectious disease, including but not limited to chronic renal infection, chronic chest infection (e.g. bronchectasis), sinusitis, recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremeting cystitis) open, draining or infected skin wound, or ulcer. Serious infection(s) (such as hepatitis, pneumonia or pyelonephritis) within 3 months prior to inclusion.
  * Malignancy within the previous 5 years with the exception of basal cell carcinoma of the skin that has been treated with no evidence of recurrence.
  * Active tuberculosis or previous history of non treated or insufficiently treated tuberculosis.
* Patients with a positive intradermal tuberculosis test according to the local recommendation
* For the patients who could have been in contact with a person having tuberculosis, the inclusion will be possible under specific conditions depending of local recommendations issued in France, Denmark, Hungary, Italy, Spain.

  * Herpes zoster (shingles) infection within 2 months prior to the first infusion
  * Opportunistic infections, e.g. cytomegalovirus, Pneumocystis carinii pneumonia, aspergillosis, histoplasmosis or atypical mycobacterium infection.
* Has any of the following clinical conditions:

  * Severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, psychiatic or cerebral diseases
  * Known to be infected with human immunodeficiency virus (HIV), hepatitis B or hepatitis C
  * Known lymphoproliferative disease, including lymphoma, or signs suggestive of lymphoproliferative disease, such as lymphadenoma of unusual size and localization or splenomegaly.
  * Have received live (attenuated) vaccination during the last 30 days
  * Have been treated with a monoclonal antibody or a fusion protein except etanercept, adalimumab or any other anti TNF agent
* Leukopenia < 3,500/mm^3, Hemoglobin < 9g/dl, thrombopenia < 100,000/mm^3.
* Congestive heart failure (CHF) including medically controlled, asymptomatic CHF or unstable hemodynamic cardiac conditions.
* Scheduled surgical intervention at any time during the study.
* Multiple sclerosis or symptomatic demyelination of central nervous system.
* Subjects who have an history of drug abuse or alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infliximab 5 mg/kg
Started | 7
Completed | 1
Not Completed | 6
Not completed — Relapse | 2
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: The Number of Enthesitis Between Week 4 and Week 12 Evaluated Using Power Doppler Ultrasonography (PDUS) and Proprietary Software.
Description: Two measures were to be used for each enthesis evaluation. 1.) Vascularization: yes/no. 2.) Area of hyper-vascularization: mm^2 (continuous) using proprietary software. This study was terminated early due to slow recruitment. As a result, efficacy analyses were not performed.
Time Frame: 8 weeks
Measure: Number; unit: Number of Enthesitis
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 7
Number of Enthesitis | 0

ADVERSE EVENTS:
Arm/Group | Infliximab 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg (N=7)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis Generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Skin Plaque (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees not to publish or publicly present any interim results of the study without prior written consent of the sponsor. The PI further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication which report any results of the study. The sponsor shall have the right to review and comment on any presentation.